CLINICAL TRIAL: NCT04681976
Title: Effectiveness of a Telematic Dance Intervention on the Quality of Life of Older People: Randomized Clinical Trial
Brief Title: Telematic Dance Intervention on Quality of Life of Older
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Francisco Martínez Arnau, Physiotherapist, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1493554
Record Dates: First submitted 2020-12-16; First posted 2020-12-23 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Aging Well
Keywords: older; dance; muscle strenght; quality of life

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention Group participants will perform a 3-month telematic dance program based on choreographic work, 2 times per week
  Interventions: Behavioral: Telematic dance program
- Control group (No Intervention): Control group will follow their daily routine without added exercise

INTERVENTIONS:
Behavioral: Telematic dance program — Telematic dance program
  The dance program will consist of 24 sessions distributed twice a week for a total period of 3 months. Each session will include:
  A) Warm up: It will consist of analytical and global movements of increasing intensity and stretching exercises. It will also involve body awareness and motor control exercises.
  B) Choreography part: the participants must follow and learn the choreographies. Intensity ranges shall vary between low and moderate. (3-4 in Borg's Modified Scale (0-10)).
  C) Cool down: It will consist of global movements of decreasing intensity, stretching, breathing, and relaxing exercises.
  Arms: Intervention group

SUMMARY:
The aim of this study is to analyse the effectiveness of a telematic dance intervention on the quality of life of older people.

This project is a controlled, randomized clinical trial. 54 people (Intervention Group, n=27; Control Group, n=27) between the ages of 60-80 will participate in the study.

Intervention Group participants will perform a 3-month telematic dance program based on choreographic work. The participants shall be measured 3 times, at baseline, post-intervention, and at 6-month post-intervention follow-up. Aside from the quality of life, variables of balance, risk of falling, number of falls, level of physical activity, mood, functionality, comorbidity, and quadriceps strength will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60-80.
* Owning a device that can connect to internet to visualize videos and do videocalls, in case a session to resolve doubts is necessary.

Exclusion Criteria:

* Subjects with degenerative or cognitive pathologies
* Subjects with severe visual deficiencies.
* Subjects with any acute pain.
* Subjects with inability to stand.
* Subjects with any medical contraindication to exercise (cardiovascular risk factors).
* Subjects incapable of managing telematic devices to follow the sessions.
* Subjects who refuse to sign the informed consent.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Changes in quality of Life | 0-3 months
  Changes produced by a 3-month telematic dance program related to quality of life (EuroQol 5 Dimensions - 3 levels Index, 0 to 1 point, higher values = better outcome).

SECONDARY OUTCOMES:
Adherence | 0-3 months
  Measurement of adherence (expressed in % of assistance to the 24 sessions) to the 3-month telematic dance program.
Body composition | 0-3 months
  Changes on body composition (measured by bioimpedance in %) generated by 3-month telematic dance program
Balance | 0-3 months
  Changes on balance produced by a 3-month dance program measured by Timed Up and Go Test (measured in seconds) and one single leg stance test (measured in seconds).
Fear of falling | 0-3 months
  Changes on fear of falling measured by Falls Efficacy Scale-International (16 items measured by 4 point Lickert scale; 1= not worried, 4= very worried, (0-64)), and number of falls (retractive, 3 previous months and prospective, 3 following months).
Level of physical activity | 0-3-6 months
  Changes in the level of physical activity measured by the International Physical Activity Questionnaire (IPAQ) (expressed in minutes) produced by a 3-month telematic dance program
Mood | 0-3-6 months
  Changes in mood measured by the Mood Evaluation Scale (16 items measured in Likert scales (0-10)) produced by a 3-month telematic dance program.
Functionality | 0-3 months
  Changes in functionality and independence measured by Barthel Index (0 to 100 points, < 60 dependence, higher values = better outcome) produced by a 3-month telematic dance program.
Knee extension isometric strength | 0-3 months
  Changes produced in knee extension isometric strength measured with dynamometer (N) by a 3-month telematic dance program

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Martínez-Arnau, PhD, Principal Investigator — Universitat de Valencia
Locations (1):
- University of Valencia - Faculty of Physiotherapy, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No